CLINICAL TRIAL: NCT04915378
Title: Does Hypoxia-altitude Testing at Lowland Predict Altitude Related Adverse Health Effects in COPD Patients Traveling to 3100m?
Brief Title: Hypoxia-altitude Testing to Predict Altitude Related Adverse Health Effects in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine, Kyrgyz Republic (Unknown)
Responsible Party: Sponsor
Other Study IDs: 01-2021-SU-HAST
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Hypoxia Altitude Simulation Test; High Altitude
Keywords: Hypoxia altitude simulation test (HAST); Chronic obstructive pulmonary disease; Mountain Sickness; Altitude-related adverse health effects (ARAHE)
MeSH Terms: conditions — Altitude Sickness; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: hypoxia altitude simulation test (HAST) at 760m — Normobaric hypoxia at a FiO2 of 15.1% will be generated by the Everest Summit II altitude generator (Hypoxico Altitude Training Systems, Bickenbach, Germany) and delivered to the patients face via tubes and a tightly fitted mask. Patients will be seated comfortably in a chair and fitted with a full-face mask equipped with a one-way valve. After a baseline period of quiet rest of 5-10 min with ambient air breathing and installation of equipment, patients will breath the hypoxic air mixture via a tightly fitted facial mask. They will be monitored with a finger-tip pulseoximetry to continuously assess SpO2 and heart rate. After at least 15' and steady-state values of the SpO2 (±1%) for at least 5' arterial blood gases will be drawn from a radial artery and immediately analyzed (RapidPoint 500, Siemens, Zürich, Switzerland).
Procedure: High Altitude (3100m) — High Altitude (3100m) exposure for 2 days

SUMMARY:
The predictive value of the hypoxia altitude simulation test (HAST) or other baseline values to predict altitude-related adverse health effects (ARAHE) is not established. To address this gap, the main goals of this investigation will be 1) to evaluate the diagnostic accuracy of the HAST in identifying individuals that will experience ARAHE during altitude travel and 2) to establish prediction models incorporating other commonly assessed clinical characteristics either alone or in combination with the HAST as predictors of ARAHE in altitude travelers.

Hypotheses: In lowlanders with COPD, a PaO2 <6.6 kPa or another cutoff of PaO2 or SpO2 at the end of the HAST, at rest or during exertion and/or clinical variables including symptoms, pulmonary function indices, 6-min walk distance (6MWD), either alone or combined to a multivariable model, will predict ARAHE during a sojourn of 2 days at 3100m with accuracy greater than chance

DETAILED DESCRIPTION:
Altitude or air travel has become increasingly popular for recreational and professional reasons. Chronic obstructive pulmonary disease (COPD) affects up to 12% of adults worldwide and is associated with progressive hypoxemia, especially during exercise, due to respiratory mechanical constraints, airway obstruction and increasing pulmonary hypertension (PH). COPD patients are at increased risk of ARAHE including acute mountain sickness (AMS) and severe hypoxemia. Factors assessed at lowland that would predict ARAHE of COPD patients exposed to a hypobaric hypoxic environment at altitude or during air travel would be highly warranted. During the HAST COPD-patients are exposed to an inspiratory oxygen fraction (FiO2) of 15.1% corresponding to an altitude of ≈ 2500m and this test was designed to predict deoxygenation at altitude. The predictive value of the HAST or other baseline values to predict ARAHE is not established. To address this gap, the main goals of this investigation will be 1) to evaluate the diagnostic accuracy of the HAST in identifying individuals that will experience ARAHE during altitude travel and 2) to establish prediction models incorporating other commonly assessed clinical characteristics either alone or in combination with the HAST as predictors of ARAHE in altitude travelers.

For this diagnostic accuracy study, COPD-patients with an FEV1 40-80% predicted living < 1000 m without severe hypoxemia (SpO2, <92%), hypercapnia (PaCO2 >6 kPa) or comorbidities will be recruited to traveling to and staying for two nights at 3100 m. At 760 m, the HAST will be performed, at 760 m and 3100 m symptoms, vital signs, SpO2, pulmonary function tests, 6MWD, sleep studies will be repetitively assessed. ARAHE will be defined if one of the following present: AMS with a Lake Louise questionnaire score >4 including headache, or AMSc score ≥0.7, resting SpO2 <80% >30 min or <75% for >15 min; or exercise SpO2 <75% for >5 min accompanied by symptoms, any intercurrent illness including infections, hypertension, neurologic impairments, dyspnea or discomfort at rest requiring oxygen treatment, chest pain and/or ECG signs of cardiac ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 35-75 y, living at low altitude (<800 m).
* COPD diagnosed according to the Global Initiative for Obstructive Lung Disease (GOLD) guidelines, FEV1 40-80% predicted, pulse oximetry ≥92%, PaCO2 <6 kPa, breathing ambient air at 760 m.

Exclusion Criteria:

* COPD exacerbation, very severe COPD with hypoxemia or hypercapnia at 760 m (see above).
* Other lung disease, relevant comorbidities (such as uncontrolled cardiovascular disease, i.e., unstable arterial hypertension, coronary artery disease; previous stroke; obesity (body mass index >35 kg/m2); internal, neurologic, rheumatologic or psychiatric disease; current heavy smoking (>20 cigarettes per day).
* Renal failure and/or allergy to sulfonamides.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD-patients living in the Bishkek area (mean altitude 760m) will be recruited among patients of the outpatient clinic of the National Center for Cardiology and Internal Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
PaO2 <6.6 kPa or SpO2 < 85% during a HAST in identifying participants with ARAHE | 3 days
  Accuracy of a PaO2 <6.6 kPa during a HAST in identifying participants with ARAHE during the ascent to and stay for 2 days at 3'100 m

SECONDARY OUTCOMES:
pulse oximetry (SpO2) | 3 days
  At 760 m and 3100m
six minute walking distance | 3 days
  At 760 m and 3100m
pulmonary function | 3 days
  Spirometry and single breath carbon monoxide diffusing capacity will be measured
Nocturnal respiratory polygraphies | 2 nights
  Real-time polygraphic data and videostreams will be transmitted to a control station to allow continuous observation by an investigator. This will allow detection of ARAHE at night (in particular severe hypoxemia)
Borg Dyspnea Scale | 3 days
  Borg Scale for dyspnea from 0 to 10 (CR10) while 0 means "no dyspnea" and 10 means "highest dyspnea", to assess dyspnea at 760 m and 3100m
Lake Louise score (2018 version) | 3 days
  Which includes self-assessment of symptoms (headache, fatigue, gastrointestinal discomfort, dizziness), each rated from 0 (absent) to 3 (severe) at 760 m and 3100m.
Environmental Symptoms Questionnaire cerebral score | 3 days
  Environmental Symptoms Questionnaire cerebral score (AMSc) comprising 11 questions on symptoms rated from 0 (not at all) to 5 (extreme). The weighted sum of responses ranges from 0 to 5. At 760 m and 3100m.
Arterial blood gas analysis | 3 days
  To assess arterial partial pressure of oxygen (PaO2) at 760 m and 3100m
The Karolinska sleepiness scale | 2 nights
  Sleepiness will be assessed by the Karolinska sleepiness scale at 3200 m. This is a 9-point scale (1 = extremely alert, 3 = alert, 5 = neither alert nor sleepy, 7 = sleepy - but no difficulty remaining awake, and 9 = extremely sleepy - fighting sleep).
Blood pressure | 3 days
  At 760 m and 3100m.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof, Study Chair — University Hospital, Zürich, Switzerland; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: No